CLINICAL TRIAL: NCT06776276
Title: The Impact of Adding Tai-chi Training to Pharmacotherapy in Post Covid Insomnia: a Prospective Study.
Brief Title: A Prospective Study: Tai-chi and Post-COVID Insomnia
Acronym: insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0305339; no funding (Other: no funding)
Record Dates: First submitted 2025-01-11; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2020-09

CONDITIONS: Insomnia; COVID - 19
Keywords: Insomnia; COVID-19; Tai Chi exercises; Insomnia severity index
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post-COVID Insomnia (Active Comparator)
  Interventions: Behavioral: Tai Chi exercises
- non-COVID-19-related insomnia (No Intervention)

INTERVENTIONS:
Behavioral: Tai Chi exercises — Tai-chi (TC) is a kind of CAM Qigong exercises, is a type of classic Chinese martial arts. It entails deliberate, slow-motion physical movements that are done alongside inward concentration, awareness of breathing, and the inherent power or energy in the body. It promotes general purposes of health and spirituality. It is generally accessible and offered to older people in public places.
  Arms: Post-COVID Insomnia

SUMMARY:
The goal of this study is to see if Tai-Chi exercises (a type of Chinese martial arts) can help people suffering from insomnia after COVID-19 when added with cognitive-behavioral therapy (CBT) and drugs compared to CBT and drugs alone. All participants will receive education on sleep hygiene practices, and the principles of cognitive behavioral therapy (CBT). If these approaches were insufficient, they will be given sleep aids, primarily Z-drugs.

All study subjects engaged in a simple Tai Chi training program for two weeks. The Tai Chi training consisted of a series of gentle physical exercises that incorporated elements of meditation, body awareness, imagery, and abdominal breathing.

A professional instructor conducted two training sessions for both patients and controls, ensuring that participants could perform the exercises independently at home during the last hour before sleep. Each session lasted twenty minutes, to be done daily. Participants were given a checklist documenting their sleep and exercise diary to confirm adherence for at least five days each week. After the two-week period, all participants are reassessed using the Insomnia severity index.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infections confirmed by PCR (polymerase chain reaction)
* Over the age of 18 years

Exclusion Criteria:

* Below the age of 18 years
* Severely ill patients
* Patients with chronic respiratory complications
* Individuals with pre-existing and ongoing depression or anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | from enrollment to the end of treatment at 2 weeks follow up timestamp
  The ISI measures the frequency of various insomnia symptoms, including prolonged sleep latency, difficulty maintain sleep, early awakening, satisfaction with sleep, interference with the daily activities, if it is noticed by others and if it is causing distress. Each of the seven items is rated on a 5-point Likert scale, ranging from 0 (no problem) to 4 (very severe problem), resulting in a total score that can range from 0 to 28.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Osypiuk K, Thompson E, Wayne PM. Can Tai Chi and Qigong Postures Shape Our Mood? Toward an Embodied Cognition Framework for Mind-Body Research. Front Hum Neurosci. 2018 May 1;12:174. doi: 10.3389/fnhum.2018.00174. eCollection 2018. PMID 29765313
- [Background] Chan SH, Ng SM, Yu CH, Chan CM, Wang SM, Chan WC. The effects of an integrated mindfulness-based tai chi chuan programme on sleep disturbance among community-dwelling elderly people: protocol for a randomized controlled trial. Trials. 2022 Sep 24;23(1):808. doi: 10.1186/s13063-022-06737-4. PMID 36153623
- [Background] Tong Y, Chai L, Lei S, Liu M, Yang L. Effects of Tai Chi on Self-Efficacy: A Systematic Review. Evid Based Complement Alternat Med. 2018 Aug 15;2018:1701372. doi: 10.1155/2018/1701372. eCollection 2018. PMID 30186352